CLINICAL TRIAL: NCT00794157
Title: A 12-week Treatment, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Indacaterol (150 and 300 µg Once Daily [od]) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Confirmatory Study of Indacaterol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B1302
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; chronic obstructive pulmonary disease; indacaterol; long acting β2-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Indacaterol 150 µg (Experimental): Patients received indacaterol 150 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg capsules
- Indacaterol 300 µg (Experimental): Patients received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg capsules
- Placebo (Placebo Comparator): Patients received placebo delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Indacaterol 150 μg capsules — Indacaterol was supplied in powder filled capsules with a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 150 µg
Drug: Indacaterol 300 μg capsules — Indacaterol was supplied in powder filled capsules with a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 300 µg
Drug: Placebo capsules — Placebo was supplied in powder filled capsules with a single dose dry powder inhaler (SDDPI).
  Arms: Placebo

SUMMARY:
This study was designed to provide pivotal confirmation of efficacy and safety data for 2 doses of indacaterol (150 and 300 µg once daily [od]) in patients with moderate to severe chronic obstructive pulmonary disease (COPD). Data from this study will be used for the registration of indacaterol in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-to-severe chronic obstructive pulmonary disease (COPD), as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines and:

  1. Smoking history of at least 20 pack-years.
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value.
  3. Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%.

Exclusion Criteria:

* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to screening or during the 14 day run-in period prior to randomization.
* Patients requiring long-term oxygen therapy (> 15 hours a day) for chronic hypoxemia.
* Patients who have had a respiratory tract infection within 6 weeks prior to screening.
* Patients with concomitant pulmonary disease.
* Patients with a history of asthma.
* Patients with diabetes Type I or uncontrolled diabetes Type II.
* Any patient with lung cancer or a history of lung cancer.
* Any patient with active cancer or a history of cancer with less than 5 years disease-free survival time.
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at screening or randomization is prolonged.
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period.
* Patients unable to successfully use a dry powder inhaler device or perform spirometry measurements.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- Hong Kong (2):
  - Novartis Investigator Site, Hong Kong
  - Novartis Investigator Site, New Territories
- India (7):
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigator Site, Bangalore
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigator Site, India
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Center, Panjim
- Japan (34):
  - Novartis Investigative Site, Asahikawa
  - Novartis Investigative Site, Bunkyō City
  - Novartis Investigator Site, Gifu
  - Novartis Investigator Site, Himeji
  - Novartis Investigator Site, Hiroshima
  - Novartis Investigator Site, Iwata
  - Novartis Investigator Site, Kanazawa
  - Novartis Investigative site, Kawasaki
  - Novartis Investigator Site, Kishiwada
  - Novartis Investigator Site, Kitakyushu
  - Novartis Investigator Site, Kochi
  - Novartis Investigator Site, Koga
  - Novartis Investigative Site, Kurume
  - Novartis Investigator Site, Kyoto
  - Novartis Investigative Site, Maebashi
  - Novartis Investigator Site, Matsusaka
  - Novartis Investigative Site, Morioka
  - Novartis Investigator Site, Nagaoka
  - Novartis Investigator Site, Nagoya
  - Novartis Investigative Site, Noda
  - Novartis Investigative Site, Obihiro
  - Novartis Investigator Site, Sakai
  - Novartis Investigative Site, Sapporo
  - Novartis Investigator Site, Sendai
  - Novartis Investigator Site, Seto
  - Novartis Investigator Site, Tenri
  - Novartis Investigative site, Tokyo
  - Novartis Investigator Site, Toyonaka
  - Novartis Investigator Site, Ube
  - Novartis Investigator Site, Wakayama
  - Novartis Investigator Site, Yabu
  - Novartis Investigator Site, Yanagawa
  - Novartis Investigator Site, Yokkaichi
  - Novartis Investigative Site, Yokohama
- Novartis Investigator Site, Singapore, Singapore
- South Korea (6):
  - Novartis Investigator Site, Daegu
  - Novartis Investigator Site, Junggu
  - Novartis Investigative Site, Kangwon-Do
  - Novartis Investigator Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigator Site, Seoul
- Taiwan (10):
  - Novartis Investigator Site, Chiayi City
  - Novartis Investigator Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taichung
  - Novartis Investigator Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigator Site, Taipei
  - Novartis Investigator Site, Taipei County
  - Novartis Investigator Site, Xindian District

REFERENCES:
- [Derived] To Y, Kinoshita M, Lee SH, Hang LW, Ichinose M, Fukuchi Y, Kitawaki T, Okino N, Prasad N, Lawrence D, Kramer B. Assessing efficacy of indacaterol in moderate and severe COPD patients: a 12-week study in an Asian population. Respir Med. 2012 Dec;106(12):1715-21. doi: 10.1016/j.rmed.2012.09.002. Epub 2012 Oct 5. PMID 23040786

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol 150 μg: Patients received indacaterol 150 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 300 μg: Patients received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Period: Overall Study
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Started | 114 | 116 | 117
Completed | 104 | 106 | 98
Not Completed | 10 | 10 | 19
Not completed — Adverse Event | 4 | 1 | 8
Not completed — Subject withdrew consent | 2 | 0 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 2
Not completed — Administrative problems | 1 | 7 | 4
Not completed — Abnormal test procedure result(s) | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo | Total
Number analyzed (Participants) | 114 | 116 | 117 | 347
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.75) | 67.1 (7.67) | 66.5 (8.74) | 66.7 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 110 | 113 | 112 | 335

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of Treatment (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 60 minutes post-dose of ipratropium during screening as covariates.
Time Frame: End of treatment (Week 12 + 1 day, Day 85)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug. The imputation technique used as last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 109 | 110 | 104
Liters | 1.34 (0.024) | 1.37 (0.023) | 1.17 (0.025)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Week 2. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 60 minutes post-dose of ipratropium during screening as covariates.
Time Frame: After Week 2 (Day 15)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 93 | 85 | 82
Liters | 1.33 (0.023) | 1.34 (0.023) | 1.17 (0.024)

3. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 4
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Week 4. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 60 minutes post-dose of ipratropium during screening as covariates.
Time Frame: After Week 4 (Day 29)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 81 | 82 | 80
Liters | 1.32 (0.024) | 1.33 (0.022) | 1.18 (0.024)

4. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 8
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Week 8. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 60 minutes post-dose of ipratropium during screening as covariates.
Time Frame: After Week 8 (Day 57)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 81 | 79 | 71
Liters | 1.30 (0.029) | 1.32 (0.027) | 1.14 (0.030)

5. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12 (Day 84)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 50 and 15 minutes pre-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 60 minutes post-dose of ipratropium during screening as covariates.
Time Frame: Prior to last dose at Week 12 (Day 84)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Number analyzed (Participants) | 81 | 79 | 70
Liters | 1.34 (0.032) | 1.34 (0.030) | 1.13 (0.031)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population.
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/114 | 2/116 | 6/117
Other Adverse Events (participants affected / at risk) | 24/114 | 26/116 | 26/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=114) | Indacaterol 300 μg (N=116) | Placebo (N=117)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Concomitant disease progression (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=114) | Indacaterol 300 μg (N=116) | Placebo (N=117)
Nasopharyngitis (Infections and infestations) | 10 | 8 | 11
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.